CLINICAL TRIAL: NCT06963775
Title: Assessment of Traumatic Brain Injury Using Transcranial Magnetic Stimulated Evoked Potentials (TMS-EEG)
Brief Title: Assessment of Traumatic Brain Injury Using Transcranial Magnetic Stimulated Evoked Potentials
Acronym: (TMS-EEG)
Status: Not yet recruiting | Type: Observational
Sponsor: Ramon Diaz-Arrastia (Other)
Collaborators: QuantalX Neuroscience (Industry)
Responsible Party: Sponsor-Investigator, Ramon Diaz-Arrastia, Presidential Professor & Director of Clinical Traumatic Brain Injury Research Initiative, University of Pennsylvania Perelman School of Medicine, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Other Study IDs: 855370
Record Dates: First submitted 2025-03-07; First posted 2025-05-09 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Traumatic Brain Injury; TMS-EEG; neurological disorders
MeSH Terms: conditions — Brain Injuries, Traumatic; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Traumatic Brain Injury (Acute, Subacute, Chronic)
  Interventions: Device: Delphi-MD device (QuantalX Neuroscience Ltd., Saba Israel)
- Healthy Control
  Interventions: Device: Delphi-MD device (QuantalX Neuroscience Ltd., Saba Israel)

INTERVENTIONS:
Device: Delphi-MD device (QuantalX Neuroscience Ltd., Saba Israel) — Delphi-MD utilizes the use of transcranial magnetic stimulation evoked electroencephalography (TMS-EEG) for diagnostic purposes in a wide range of neurological disorders. Delphi-MD includes a magnetic stimulator and coil, an EEG amplifier and electrode cap and software for the acquisition and analysis of the data.
  Delphi-MD stimulation protocol includes low intensities (sub motor thresholds) and frequencies over six stimulation sites (bilateral primary motor cortex, and bilateral dorsolateral prefrontal cortex).

SUMMARY:
Patients evaluated at Penn Presbyterian Medical Center for traumatic brain injury (TBI), who sign the informed consent, will undergo assessment of electrophysiologic potentials evoked by transcranial magnetic stimulation (TMS), using the Delphi-MD device (QuantalX Neuroscience Ltd., Saba Israel).

ELIGIBILITY:
Inclusion Criteria for Traumatic Brain Injury (Acute, Subacute, Chronic) group:

1. Age 18 years and older
2. Evidence of mechanical energy impacting the head or inertial forces affecting the head
3. Either (A) or (B):

   1. Trauma-related abnormality on CT scan on admission
   2. If CT normal, documented/verified TBI based on evidence of either loss of consciousness, post-traumatic amnesia, confusion, or post-traumatic symptoms.

Exclusion Criteria for Traumatic Brain Injury (Acute, Subacute, Chronic) group:

1. History of disabling pre-existing neurologic disease (Such as epilepsy, brain tumors, meningitis, cerebral palsy, encephalitis, brain abscesses, vascular malformations, cerebrovascular disease, Alzheimer's disease, multiple sclerosis, or HIV-encephalitis)
2. History of premorbid disabling condition that interfere with outcome assessments
3. Bilaterally absent pupillary responses
4. Penetrating traumatic brain injury
5. Prisoners or patients in police custody
6. Pregnancy
7. Subjects with magnetic-sensitive devices implanted in their head or within 12 in. (30 cm) of the coil/probe (examples: cochlear implants, deep brain stimulators, vagus nerve stimulators, other implanted electrodes/stimulators, aneurysm clips or coils, stents and bullet fragments).

Inclusion Criteria for Healthy Control group:

1. Age 18 years and older
2. No history of TBI in the past 12 months

Exclusion Criteria for Healthy Control group:

1. History of disabling pre-existing neurologic disease (Such as epilepsy, brain tumors, meningitis, cerebral palsy, encephalitis, brain abscesses, vascular malformations, cerebrovascular disease, Alzheimer's disease, multiple sclerosis, or HIV-encephalitis)
2. History of premorbid disabling condition that interfere with outcome assessments
3. Prisoners or patients in police custody
4. Pregnancy
5. Subjects with magnetic-sensitive devices implanted in their head or within 12 in. (30 cm) of the coil/probe (examples: cochlear implants, deep brain stimulators, vagus nerve stimulators, other implanted electrodes/stimulators, aneurysm clips or coils, stents and bullet fragments).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll up to 145 patients with a traumatic brain injury diagnosis evaluated at University of Pennsylvania Health System over 5 years. We will also evaluate up to 70 uninjured healthy controls, matched by age and gender to TBI participants.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
1. Differentiate between healthy controls and TBI participants in measured outputs of the DELPHI-MD device (WFA, STP, EPD, LPD, and Connectivity) | Day 1
  1. WFA (Waveform Adherence)
  2. STP (short-term plasticity)
  3. EPD (Early Phase Deflection)
  4. LPD (Late Phase Deflection)
  5. Connectivity (these are all in arbitrary units)
2. Correlate DELPHI-MD outputs with neural deficits identified through patient reported and clinician reported outcome measures | Day 1
  For single timepoint (day 1).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy-Lamdan O, Zifman N, Sasson E, Efrati S, Hack DC, Tanne D, Dolev I, Fogel H. Evaluation of White Matter Integrity Utilizing the DELPHI (TMS-EEG) System. Front Neurosci. 2020 Dec 21;14:589107. doi: 10.3389/fnins.2020.589107. eCollection 2020. PMID 33408607
- [Background] Fogel H, Levy-Lamdan O, Zifman N, Hiller T, Efrati S, Suzin G, Hack DC, Dolev I, Tanne D. Brain Network Integrity Changes in Subjective Cognitive Decline: A Possible Physiological Biomarker of Dementia. Front Neurol. 2021 Aug 30;12:699014. doi: 10.3389/fneur.2021.699014. eCollection 2021. PMID 34526957
- [Background] Zifman N, Levy-Lamdan O, Suzin G, Efrati S, Tanne D, Fogel H, Dolev I. Introducing a Novel Approach for Evaluation and Monitoring of Brain Health Across Life Span Using Direct Non-invasive Brain Network Electrophysiology. Front Aging Neurosci. 2019 Sep 9;11:248. doi: 10.3389/fnagi.2019.00248. eCollection 2019. PMID 31551761
- [Background] Zifman N, Levy-Lamdan O, Hiller T, Thaler A, Dolev I, Mirelman A, Fogel H, Hallett M, Maidan I. TMS-evoked potentials unveil occipital network involvement in patients diagnosed with Parkinson's disease within 5 years of inclusion. NPJ Parkinsons Dis. 2024 Sep 30;10(1):182. doi: 10.1038/s41531-024-00793-0. PMID 39349492
- [Background] Lassman S, Zifman N, Fogel H, Hassin-Baer S, Anis S. TMS-evoked potentials provide novel neurophysiological features of Tourette syndrome. Parkinsonism Relat Disord. 2025 Jan;130:107217. doi: 10.1016/j.parkreldis.2024.107217. Epub 2024 Nov 22. PMID 39612660
- [Background] Maidan I, Zifman N, Hausdorff JM, Giladi N, Levy-Lamdan O, Mirelman A. A multimodal approach using TMS and EEG reveals neurophysiological changes in Parkinson's disease. Parkinsonism Relat Disord. 2021 Aug;89:28-33. doi: 10.1016/j.parkreldis.2021.06.018. Epub 2021 Jun 29. PMID 34216938
- See also: Study device — https://quantalx.com/delphi-md/